CLINICAL TRIAL: NCT02951975
Title: Multicentre Longitudinal Study of the Prescription of Ozurdex® in Patients With Non-infectious Uveitis Affecting the Posterior Segment of the Eye
Brief Title: Ozurdex® in Patients With Non-infectious Uveitis Affecting the Posterior Segment of the Eye
Acronym: Louvre 2
Status: Terminated | Type: Observational
Why Stopped: Business decision to stop the program.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-EAME-EYE-0368
Record Dates: First submitted 2016-10-31; First posted 2016-11-01 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Non-infectious Uveitis
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OZURDEX®: Patients prescribed dexamethasone intravitreal implant (OZURDEX®) in clinical practice for the treatment of non-infectious uveitis affecting the posterior segment of the eye.
  Interventions: Drug: dexamethasone intravitreal implant

INTERVENTIONS:
Drug: dexamethasone intravitreal implant — Dexamethasone intravitreal implant (OZURDEX®) as prescribed in clinical practice.
  Other Names: OZURDEX®

SUMMARY:
This observational study will evaluate the safety, efficacy, characteristics of patients, characteristics of physicians and quality of life in patients who are prescribed OZURDEX® as treatment for non-infectious uveitis of the posterior segment of the eye in France.

ELIGIBILITY:
Inclusion Criteria:

-Patient with non-infectious uveitis affecting the posterior segment of the eye.

Exclusion Criteria:

-Patient not residing in metropolitan France.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with OZURDEX® in clinical practice.
Sampling Method: Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Best Corrected Visual Acuity (BCVA) ≥15 Letters | 2 Months

SECONDARY OUTCOMES:
Percentage of Participants with a Gain (Improvement) in BCVA of at Least 15 Letters from Baseline | Baseline, Months 6 and 18
Change from Baseline in BCVA | Baseline, Months 2, 6 and 18
Change from Baseline in Vitreous Haze Score Using a 5-Point Scale | Baseline and Months 2, 6 and 18
Change from Baseline in Macular Thickness | Baseline, Months 2, 6 and 18
Percentage of Participants Categorized by Comorbidities (Diseases Associated with Inflammation, Other Ophthalmic Diseases, General Comorbidities) | 18 Months
Change from Baseline in the National Eye Institute-Visual Function Questionnaire-25 (NEI-VFQ25) Score Using a 25 Item Questionnaire | Baseline, Months 2 and 18
Number of Repeat Treatments with OZURDEX® and Other Drugs | 18 Months
Time Between Repeat Treatments with OZURDEX® and Other Drugs | 18 Months
Percentage of Participants with Adverse Events (AEs) | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Mesnard, Study Director — Allergan
Locations (21):
- France (21):
  - CHU Amiens, Amiens
  - IOP Institut Ophtalmologique de Picardie, Amiens
  - Centre Rétine Gallien, Bordeaux
  - Hopital Pellegrin, Bordeaux
  - CHI de Créteil, Créteil
  - CHU Dijon, Dijon
  - Centre Pôle Vision Val d'Ouest, Écully
  - Hopital Claude Huriez, Lille
  - Hopital De La Croix Rousse, Lyon
  - Clinique Monticelli, Marseille
  - Hopital de la Timone, Marseille
  - Hopital Gui De Chauliac, Montpellier
  - SEL Ophtalliance, Nantes
  - Hopital Hotel Dieu Et Hme, Nantes
  - CHU Pasteur 2, Nice
  - Hôpital Lariboisière (AP-HP), Paris
  - GH Pitie Salpêtrière (AP-HP), Paris
  - GH Cochin St Vincent De Paul (AP-HP), Paris
  - Fondation Rothschild, Paris
  - Hopital La Milétrie, Poitiers
  - Chu Toulouse, Toulouse

REFERENCES:
- [Derived] Bodaghi B, Brezin AP, Weber M, Delcourt C, Kodjikian L, Provost A, Velard ME, Barnier-Ripet D, Pinchinat S, Dupont-Benjamin L. Real-Life Efficacy, Safety, and Use of Dexamethasone Intravitreal Implant in Posterior Segment Inflammation Due to Non-infectious Uveitis (LOUVRE 2 Study). Ophthalmol Ther. 2022 Oct;11(5):1775-1792. doi: 10.1007/s40123-022-00525-8. Epub 2022 Jul 8. PMID 35802252
- See also: More Information — http://www.allerganclinicaltrials.com